CLINICAL TRIAL: NCT05470621
Title: A Cluster Randomized Controlled Trial of an After-school Playground Intervention to Improve Children's Physical, Social, and Emotional Health: The PLAYground Project
Brief Title: A Playground Training to Improve Children's Health After-school and During Recess: The PLAYground Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00015985
Record Dates: First submitted 2022-07-18; First posted 2022-07-22 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Physical Inactivity; Social Skills; Behavior, Child
Keywords: Physical Activity; Schools
MeSH Terms: conditions — Sedentary Behavior; Social Skills; Child Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Playground Curriculum Arm (Experimental): Staff (after-school staff, recess aides, and physical education teachers) receive training to implement a playground curriculum in an after-school program; children receive a training to use the curriculum during recess
  Interventions: Behavioral: PlayOn! playground curriculum
- Program As Usual (No Intervention): Staff and students receive no training and participate in after-school programs and recess as usual

INTERVENTIONS:
Behavioral: PlayOn! playground curriculum — A staff and student training to implement a playground curriculum in after-school and recess settings
  Arms: Playground Curriculum Arm

SUMMARY:
Schools are critical settings to foster children's health. The purpose of this two-year cluster-randomized trial is to enhance both the after-school and recess settings to provide children with knowledge and skills to facilitate active and inclusive play. The primary aim of the project is to assess the impact of a playground curriculum intervention on children's physical, social, emotional, and behavioral health. The secondary aim of the project to understand the appropriateness, feasibility, fidelity, and sustainability of implementing a playground curriculum in after-school and recess settings.

DETAILED DESCRIPTION:
Physical, social, and emotional health are critical for children and predict good health later in life. Schools are essential settings to foster children's health as they provide access to the majority of children during crucial stages of development. In particular, recess and before/after school programming are critical sources of children's health and well-being, and core components of a whole school approach to health and wellness. The purpose of this two-year cluster-randomized trial is to enhance the quality of these existing settings through the integration of a playground curriculum designed to promote active and inclusive play.

Based on Social Cognitive Theory aligned with the Theory of Expanded, Extended, and Enhanced Opportunities, it is hypothesized that active and inclusive play through a playground curriculum intervention will improve enjoyment, knowledge, and self-efficacy (personal conditions), social and emotional learning (behavioral conditions), and the development of peer relationships (environmental conditions) among children, leading to increased physical activity and reduced behavioral incidents. The implementation (appropriateness, feasibility, fidelity, and sustainability) of the playground curriculum intervention to improve children's health will be assessed as a secondary outcome.

Participants will be recruited from elementary schools in Mesa Public Schools (Arizona) that offer after-school programming (N=14). The intervention includes the delivery of a curriculum aimed at providing students with knowledge and skills to initiate activities using playground structures. Trainings will be delivered to staff (after-school staff, recess aides, and Physical Education teachers) and students in the after-school setting. Students attending the after-school program will become Play Leaders to transfer the knowledge and skills they learn from PlayOn! to the recess setting.

The impact of the playground curriculum intervention on children's physical, social, emotional, and behavioral health after school and during recess will be measured using surveys, observations, interviews, physical activity devices, and de-identified school behavioral information. Data will be collected at all 14 school sites each fall and spring semester. In year one, seven schools will receive the intervention. Schools will be stratified to either the intervention or control group by Title 1 status - an indicator of school-level income. In year two, the seven control schools will receive the intervention to allow all schools the opportunity to benefit from the project.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled an after-school program in Mesa Public Schools

Exclusion Criteria:

* Students in grades kindergarten or first grade will be excluded due to their young age.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 294 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Mean change in accelerometer-derived physical activity from baseline to six months | Baseline (month 0) and Post-intervention (approximately 6 months)
  Accelerometer counts of sedentary, light-, and moderate-to-vigorous physical activity levels will be segmented and processed separately to determine physical activity during recess, during school, during after-school programming, out of school, and on weekends.
Mean change in accelerometer-derived physical activity from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  Accelerometer counts of sedentary, light-, and moderate-to-vigorous physical activity levels will be segmented and processed separately to determine physical activity during recess, during school, during after-school programming, out of school, and on weekends.
Mean change in accelerometer-derived physical activity from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  Accelerometer counts of sedentary, light-, and moderate-to-vigorous physical activity levels will be segmented and processed separately to determine physical activity during recess, during school, during after-school programming, out of school, and on weekends.
Mean change in student-reported personal (emotional) health from baseline to 6 months | Baseline (month 0) and Post-intervention (approximately 6 months)
  Child-reported personal health (enjoyment, knowledge, and self-efficacy) will be collected through questionnaire with Discrete Emotions in Physical Education Scale (DEPES).
Mean change in student-reported personal (self-efficacy) health from baseline to 6 months | Baseline (month 0) and Post-intervention (approximately 6 months)
  Child-reported personal health (enjoyment, knowledge, and self-efficacy) will be collected through questionnaire with Metacognitive Process in Physical Education Questionnaire.
Mean change in student-reported personal (social) health from baseline to 6 months | Baseline (month 0) and Post-intervention (approximately 6 months)
  Child-reported personal health (enjoyment, knowledge, and self-efficacy) will be collected through questionnaire with Saunders psychosocial influences on physical activity scale.
Mean change in student-reported environmental health from baseline to 6 months | Baseline (month 0) and Post-intervention (approximately 6 months)
  Child-reported environmental health (peer relationships) will be collected through questionnaire with the ECLS-K peer relationship scale.
Mean change in student-reported behavioral health from baseline to 6 months | Baseline (month 0) and Post-intervention (approximately 6 months)
  Child-reported behavioral health (social and emotional learning) will be collected through questionnaire with the Social and Emotional Learning module of the California Healthy Kids Survey.
Mean change in student-reported personal (emotional) health from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  Child-reported personal health indicators (enjoyment, knowledge, and self-efficacy) will be collected through questionnaire with Discrete Emotions in Physical Education Scale (DEPES).
Mean change in student-reported personal (self-efficacy) health from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  Child-reported personal health indicators (enjoyment, knowledge, and self-efficacy) will be collected through questionnaire with Metacognitive Process in Physical Education Questionnaire.
Mean change in student-reported personal (social) health from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  Child-reported personal health indicators (enjoyment, knowledge, and self-efficacy) will be collected through questionnaire with Saunders psychosocial influences on physical activity scale.
Mean change in student-reported environmental health from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  Child-reported environmental health (peer relationships) will be collected through questionnaire with the ECLS-K peer relationship scale.
Mean change in student-reported behavioral health from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  Child-reported behavioral health (social and emotional learning) will be collected through questionnaire with the Social and Emotional Learning module of the California Healthy Kids Survey.
Mean change in student-reported personal (emotional) health from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  Child-reported personal health indicators (enjoyment, knowledge, and self-efficacy) collected through questionnaire with Discrete Emotions in Physical Education Scale (DEPES).
Mean change in student-reported personal (self-efficacy) health from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  Child-reported personal health indicators (enjoyment, knowledge, and self-efficacy) collected through questionnaire with Metacognitive Process in Physical Education Questionnaire.
Mean change in student-reported personal (social) health from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  Child-reported personal health indicators (enjoyment, knowledge, and self-efficacy) collected through questionnaire with Saunders psychosocial influences on physical activity scale.
Mean change in student-reported environmental health from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  Child-reported environmental health (peer relationships) will be collected through questionnaire with the ECLS-K peer relationship scale.
Mean change in student-reported behavioral health from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  Child-reported behavioral health (social and emotional learning) will be collected through questionnaire with the Social and Emotional Learning module of the California Healthy Kids Survey.
Change in number of school-reported behavioral incidents from baseline to 6 months | Baseline (month 0) and Post-intervention (approximately 6 months)
  School-reported number of children referred to administrators for behavioral incidents
Change in number of school-reported behavioral incidents from baseline to 12 months | Baseline (month 0) and Post-intervention (approximately 12 months)
  School-reported number of children referred to administrators for behavioral incidents
Change in number of school-reported behavioral incidents from baseline to 18 months | Baseline (month 0) and Post-intervention (approximately 18 months)
  School-reported number of children referred to administrators for behavioral incidents

SECONDARY OUTCOMES:
Mean perceived implementation appropriateness | Post-intervention (approximately 6 months)
  Staff-reported appropriateness and feasibility of intervention collected through questionnaire with Intervention Appropriateness Measure (IAM).
Mean perceived implementation feasibility | Post-intervention (approximately 6 months)
  Staff-reported appropriateness and feasibility of intervention collected through questionnaire with Feasibility of Intervention Measure (FIM).
Mean observed implementation fidelity | Monthly post-intervention through end of school year
  Researcher-reported fidelity of intervention (adherence, exposure/dose, quality of delivery, component differentiation, and participant involvement) collected using researcher-developed protocol for monthly systematic observations.
Mean observed implementation sustainability | Post-intervention (approximately 12 months)
  Researcher-reported fidelity of intervention (adherence, exposure/dose, quality of delivery, component differentiation, and participant involvement) collected using researcher-developed protocol for monthly systematic observations.
Mean observed implementation sustainability | Post-intervention (approximately 18 months)
  Researcher-reported fidelity of intervention (adherence, exposure/dose, quality of delivery, component differentiation, and participant involvement) collected using researcher-developed protocol for monthly systematic observations.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Poulos, PhD, Principal Investigator — Assistant Professor, College of Health Solutions, Arizona State University; Pamela Kulinna, PhD, Principal Investigator — Professor, Mary Lou Fulton Teachers College, Arizona State University
Locations (1):
- Mesa Public Schools, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be de-identified and available
Supporting Information: Study Protocol
Time Frame: Data will become available 6 months after publication and remain available as stored in repository
Access Criteria: A link to an open-access data repository will be included in all publications. Interested parties can also contact the principal investigators of the study for data access.

REFERENCES:
- [Background] Simonton KL, Garn AC, Mercier KJ. Expanding the Discrete Emotions in Physical Education Scale (DEPES): Evaluating Emotions With Behavior and Learning. Res Q Exerc Sport. 2023 Mar;94(1):35-44. doi: 10.1080/02701367.2021.1935434. Epub 2021 Dec 14. PMID 34904920
- [Background] Saunders RP, Pate RR, Felton G, Dowda M, Weinrich MC, Ward DS, Parsons MA, Baranowski T. Development of questionnaires to measure psychosocial influences on children's physical activity. Prev Med. 1997 Mar-Apr;26(2):241-7. doi: 10.1006/pmed.1996.0134. PMID 9085394
- [Background] Jackson SL, Cunningham SA. Social Competence and Obesity in Elementary School. Am J Public Health. 2015 Jan;105(1):153-158. doi: 10.2105/AJPH.2014.302208. PMID 25393191
- [Derived] Poulos A, Kulinna PH. A cluster randomized controlled trial of an after-school playground curriculum intervention to improve children's physical, social, and emotional health: study protocol for the PLAYground project. BMC Public Health. 2022 Sep 1;22(1):1658. doi: 10.1186/s12889-022-13991-3. PMID 36050657
- See also: WestEd, California Department of Education. Using CALSCHLS to assess social-emotional learning and health [Internet]. San Francisco, CA: WestEd; 2015. — https://data.calschls.org/resources/CalSCHLS_AssessSELH.pdf

DOCUMENTS (3):
  • Study Protocol (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT05470621/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT05470621/SAP_001.pdf
  • Informed Consent Form (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT05470621/ICF_002.pdf